CLINICAL TRIAL: NCT01416142
Title: A Study to Evaluate the Product Performance of the PureVision®2 HD Contact Lens
Brief Title: A Study to Evaluate the Product Performance of the PureVision®2 High Definition (HD) Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 701E
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Results first posted 2013-12-25 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-11

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Eyeglasses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spectacles (Active Comparator): The subject's habitual spectacles (updated or confirmed as correct within the last 2 years)
  Interventions: Device: Spectacles
- PureVision2 HD contact lenses (Experimental): Currently marketed Bausch + Lomb PureVision2 HD contact lenses
  Interventions: Device: PureVision2 HD contact lenses

INTERVENTIONS:
Device: PureVision2 HD contact lenses — Lenses to be worn through 1/2 of an HD movie. Following the movie, all subjects were to wear the dispensed contact lenses on a daily wear basis for approximately one week.
  Arms: PureVision2 HD contact lenses
Device: Spectacles — Spectacles to be worn throughout 1/2 of an HD movie.
  Arms: Spectacles

SUMMARY:
The objective of this study is to evaluate the product performance of PureVision2 HD contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Have physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings
* Subjects must be myopic or hyperopic and require lens correction in each eye
* Subjects must own a pair of spectacles and the spectacle prescription must have been updated or confirmed as correct within the last 2 years.

Exclusion Criteria:

* Any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.
* Any systemic disease affecting ocular health.
* Using any systemic or topical medications that will affect ocular physiology or lens performance.
* Allergic to any component in the Biotrue multi-purpose solution

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bev Barna, CCRA, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Inc., Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant was enrolled on 7/6/2011 and last participant exited the study 8/21/2011. Participants were enrolled from 4 ophthalmology sites in the US. Study visit 1 was the screening visit, visit 2 took place in a movie theatre and visit 3 was 1 week follow-up visit.
Pre-assignment Details: 63 eligible participants were enrolled in the crossover design study, 62 participants completed the study.
Groups:
- PureVision2 HD:Spectacles: Participants:crossed over from PureVision2 HD contact lenses to spectacle wear during the movie intermission.
- Spectacles:PureVision2 HD: Participants crossed over from spectacle wear to PureVision2 HD contact lenses during the movie intermission.
- PureVision2 HD: Following the movie participants wore PureVision2 HD lenses on a daily wear basis for one week.
Period: Cross Over at Movie Intermission
Arm/Group | PureVision2 HD:Spectacles | Spectacles:PureVision2 HD | PureVision2 HD
Started | 32 | 31 | 0
Completed | 32 | 31 | 0
Not Completed | 0 | 0 | 0
Period: PureVision2 HD
Arm/Group | PureVision2 HD:Spectacles | Spectacles:PureVision2 HD | PureVision2 HD
Started | 0 | 0 | 63
Completed | 0 | 0 | 62
Not Completed | 0 | 0 | 1
Not completed — Inability to maintain lens wear | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All Eligible Baseline Participants
Groups:
- All Eligible Baseline Participants: Participants crossed over from PureVision2 HD contact lenses to spectacle wear during the movie intermission. Following the movie, all subjects were to wear the dispensed contact lenses on a daily wear basis for approximately one week.
Arm/Group | All Eligible Baseline Participants
Number analyzed (Participants) | 63
Age Continuous [Mean (Standard Deviation); unit: years] | 19.5 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Visual acuity(VA) measured at the screening visit (all eligible participants) while wearing spectacles and the VA measured at the end of study (Visit 3) 1-Week wearing PureVision2 HD lenses. VA wearing spectacles vs. VA wearing PureVision2 HD Lenses, lower the number the better the VA.
Time Frame: Screening visit (Visit 1) and one week follow-up(Visit 3)
Population: Mean scores are based on the number of eyes with nonmissing logMAR VAs. All eligible, dispensed eyes while wearing spectacles vs. wearing PureVision2 lenses.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Groups:
- PureVision2 Lenses: The currently marketed Bausch + Lomb PureVision2 HD contact lenses. Bausch + Lomb Biotrue® multi-purpose solution was dispensed with the lenses. The lower the mean logMAR the better the VA.
Arm/Group | PureVision2 Lenses | Spectacles
Number analyzed (Participants) | 45 | 45
Number analyzed (Eyes) | 90 | 90
logMAR | -0.029 (0.074) | -0.043 (0.064)

2. Secondary Outcome: Preference for Test Lens
Description: Proportion of participants preferring the Test lens over their spectacles. Participants changed from Spectacles to PureVision Lenses or PureVision Lenses to spectacles during movie intermission.
Time Frame: During the movie (Visit 2)
Population: All eligible, dispensed subjects
Measure: Number; unit: participants
Groups:
- PureVision2 Lenses: The currently marketed Bausch + Lomb PureVision2 HD contact lenses. Bausch + Lomb Biotrue® multi-purpose solution was dispensed with the lenses.
- No Difference: Participants reporting no difference between the PureVision2 HD lens and spectacles
Arm/Group | PureVision2 Lenses | Spectacles | No Difference
Number analyzed (Participants) | 56 | 56 | 56
participants
  If a choice, would you prefer glasses or contacts? | 46 | 9 | 0
  Which were more comfortable to wear? | 24 | 20 | 12
  Which provided you with superior vision? | 39 | 6 | 11
  Which made the experience more enjoyable? | 36 | 5 | 15

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | PureVision2 Lenses | Spectacles
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 0/62 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other